CLINICAL TRIAL: NCT06990919
Title: Evaluation Of The Impact Of Dental Rehabilitation Under General Anesthesia On The Stress Levels Of Children And Their Parents
Brief Title: Evaluation of the Stress Levels of Children and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Didem Sakaryali Uyar, Assoc. Prof. Dr., Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KA20/82
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Stress Biomarkers; Anxiety
Keywords: Alpha-amylase; Cortisol; Dental anxiety; general anesthesia; dental treatments
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enrolled children (Other): All of the enrolled children have been followed for 1-month. Pre-operative and post-operative saliva samples have been collected from all participating children.
  Interventions: Other: Saliva collection

INTERVENTIONS:
Other: Saliva collection — Pre-operative saliva collected before the full mouth treatment under general anesthesia while, post-operative saliva collected at 1-month follow-up after general anesthesia.

SUMMARY:
The stress levels of the participating child and their parents were evaluated using saliva to measure the stress biomarkers.

DETAILED DESCRIPTION:
All of the dental treatments of the enrolled children were performed under general anesthesia. The stress biomarkers, such as alpha-amylase and cortisol levels, were measured from the participating child's saliva samples at pre-operative and post-operative. Additionally, the stress levels of the mothers were evaluated by questionnaires at the beginning of the study.

ELIGIBILITY:
Inclusion Criteria: The children

* who did not allow their dental treatments to be completed using behavioral guidance techniques in the clinical environment.
* who had no physical or psychosocial diseases were recruited Exclusion Criteria: The children
* who were unable to give a saliva sample due to increased anxiety or inadequate saliva.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
alpha-amylase | 1-month
  salivary biomarker
cortisol | 1-month
  salivary biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data presented in this study are available from the corresponding authors upon reasonable request.